CLINICAL TRIAL: NCT03115346
Title: Alignment of Treatment Preferences and Repair Type for Veterans With AAA
Brief Title: Preferences for Open Vs. Endovascular Repair for Abdominal Aortic Aneurysm
Acronym: PROVE-AAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 15-085
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized study. Sites will be randomly assigned to the intervention group - (decision aid +survey), or control group (survey only). The randomization scheme is 9:1, for complex and intermediate VA sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- decision aid (Experimental): the experimental group will receive the decision aid
  Interventions: Other: Decision aid
- control (No Intervention): the control group will only receive the survey

INTERVENTIONS:
Other: Decision aid — Decision aid for repair type for aortic abdominal aneurysms
  Arms: decision aid

SUMMARY:
This study tests the use of a decision aid for Veterans who are facing a decision about surgery for their Abdominal Aortic Aneurysm (AAA). The local site investigators (LSI) will enroll Veterans with AAA who are candidates for endovascular or open surgical repair. There are 22-24 VA Medical Centers participating in the trial. 12 sites will be randomly assigned to the intervention group, and 12 sites will be randomly assigned to the control group. Twelve Veterans will be enrolled at each site. At sites assigned to the intervention arm, Veterans will receive a decision aid with information about the two types of surgery for AAA repair, open and endovascular, and complete a survey about their preferences. Veterans at control sites will complete the same survey, but will not receive the decision aid. After their surgery, Veterans will take another survey asking about their satisfaction. The LSI will compare the results of the survey between Veterans' in the intervention and control groups to determine the effect of the decision aid on agreement between preference and repair type.

DETAILED DESCRIPTION:
This is a cluster randomized trial comparing two ways to better align Veterans' preferences and treatments for AAA: (1) a validated decision aid describing AAA repair types with a survey measuring Veterans' preference for repair type -- versus (2) the survey alone. Enrolled Veterans will be candidates for either endovascular or open repair, and be followed at VA hospitals by vascular surgery teams who regularly perform both types of repair. In Aim 1, the investigators will determine Veterans' preferences for endovascular or open repair and identify domains associated with each repair type. In Aim 2, the investigators will compare agreement between Veterans' preferences and repair type between the decision aid+survey and survey-alone groups. In Aim 3, the investigators will investigate the facilitators and barriers of implementing a decision aid in a VA surgical clinic. The investigators will identify factors associated with agreement. The investigators' findings will be reported to the National Surgery Office Vascular Surgery Advisory Board to help ensure Veterans' preferences remain at the center of AAA treatment decisions. The investigators have recruited 20 VA Medical Centers and their vascular surgery teams to participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Veteran with a > or = 5.0 cm AAA who are candidates for both open and endovascular surgical repair, with no previous AAA repair surgery

Exclusion Criteria:

* Veterans who are not candidates for both open and endovascular repair, and are less than < 5.0 cm AAA in size

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Goodney, MD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (22):
- United States (22):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Jackson C. Montgomery VA Medical Center, Muskogee, OK, Muskogee, Oklahoma
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghaffarian AA, Griffin CL, Kraiss LW, Sarfati MR, Brooke BS. Comparative effectiveness of one-stage versus two-stage basilic vein transposition arteriovenous fistulas. J Vasc Surg. 2018 Feb;67(2):529-535.e1. doi: 10.1016/j.jvs.2017.07.115. Epub 2017 Sep 21. PMID 28943003
- [Background] Mirabelli LG, Cosker RM, Kraiss LW, Griffin CL, Smith BK, Sarfati MR, Al-Dulaimi R, Brooke BS. Rapid Methods for Routine Frailty Assessment during Vascular Surgery Clinic Visits. Ann Vasc Surg. 2018 Jan;46:134-141. doi: 10.1016/j.avsg.2017.08.010. Epub 2017 Sep 6. PMID 28887242
- [Background] Perri JL, Nolan BW, Goodney PP, DeMartino RR, Brooke BS, Arya S, Conrad MF, Cronenwett JL. Factors affecting operative time and outcome of carotid endarterectomy in the Vascular Quality Initiative. J Vasc Surg. 2017 Oct;66(4):1100-1108. doi: 10.1016/j.jvs.2017.03.426. Epub 2017 Jul 14. PMID 28712813
- [Background] DeMartino RR, Brooke BS, Neal D, Beck AW, Conrad MF, Arya S, Desai S, Aziz F, Ryan P, Cronenwett JL, Kraiss LW; Vascular Quality Initiative. Development of a validated model to predict 30-day stroke and 1-year survival after carotid endarterectomy for asymptomatic stenosis using the Vascular Quality Initiative. J Vasc Surg. 2017 Aug;66(2):433-444.e2. doi: 10.1016/j.jvs.2017.03.427. Epub 2017 Jun 2. PMID 28583737
- [Background] David RA, Brooke BS, Hanson KT, Goodney PP, Genovese EA, Baril DT, Gloviczki P, DeMartino RR. Early extubation is associated with reduced length of stay and improved outcomes after elective aortic surgery in the Vascular Quality Initiative. J Vasc Surg. 2017 Jul;66(1):79-94.e14. doi: 10.1016/j.jvs.2016.12.122. Epub 2017 Mar 31. PMID 28366307
- [Background] Brooke BS, Sarfati MR, Zhang Y, Zhang Y, Presson AP, Greene TH, Kraiss LW. Cardiac Stress Testing during Workup for Abdominal Aortic Aneurysm Repair Is Not Associated with Improved Patient Outcomes. Ann Vasc Surg. 2017 Jul;42:222-230. doi: 10.1016/j.avsg.2016.10.057. Epub 2017 Mar 10. PMID 28288889
- [Background] Williams CR, Brooke BS. Effectiveness of open versus endovascular abdominal aortic aneurysm repair in population settings: A systematic review of statewide databases. Surgery. 2017 Oct;162(4):707-720. doi: 10.1016/j.surg.2017.01.014. Epub 2017 Feb 24. PMID 28242088
- [Background] Jones DW, Schermerhorn ML, Brooke BS, Conrad MF, Goodney PP, Wyers MC, Stone DH; Vascular Quality Initiative. Perioperative clopidogrel is associated with increased bleeding and blood transfusion at the time of lower extremity bypass. J Vasc Surg. 2017 Jun;65(6):1719-1728.e1. doi: 10.1016/j.jvs.2016.12.102. Epub 2017 Feb 20. PMID 28222991
- [Background] Hoel AW, Faerber AE, Moore KO, Ramkumar N, Brooke BS, Scali ST, Sedrakyan A, Goodney PP. A pilot study for long-term outcome assessment after aortic aneurysm repair using Vascular Quality Initiative data matched to Medicare claims. J Vasc Surg. 2017 Sep;66(3):751-759.e1. doi: 10.1016/j.jvs.2016.12.100. Epub 2017 Feb 17. PMID 28222989
- [Background] Goodney PP, Spangler EL, Newhall K, Brooke BS, Schanzer A, Tan TW, Beck AW, Hallett JH, MacKenzie TA, Edelen MO, Hoel AW, Rigotti NA, Farber A. Feasibility and pilot efficacy of a brief smoking cessation intervention delivered by vascular surgeons in the Vascular Physician Offer and Report (VAPOR) Trial. J Vasc Surg. 2017 Apr;65(4):1152-1160.e2. doi: 10.1016/j.jvs.2016.10.121. Epub 2017 Feb 9. PMID 28190719
- [Background] Pannucci CJ, Swistun L, MacDonald JK, Henke PK, Brooke BS. Individualized Venous Thromboembolism Risk Stratification Using the 2005 Caprini Score to Identify the Benefits and Harms of Chemoprophylaxis in Surgical Patients: A Meta-analysis. Ann Surg. 2017 Jun;265(6):1094-1103. doi: 10.1097/SLA.0000000000002126. PMID 28106607
- [Background] Martin LA, Finlayson SRG, Brooke BS. Patient Preparation for Transitions of Surgical Care: Is Failing to Prepare Surgical Patients Preparing Them to Fail? World J Surg. 2017 Jun;41(6):1447-1453. doi: 10.1007/s00268-017-3884-z. PMID 28101609
- [Background] Bartline PB, Suckow BD, Brooke BS, Kraiss LW, Mueller MT. Outcomes in Critical Limb Ischemia Compared by Distance from Referral Center. Ann Vasc Surg. 2017 Jan;38:122-129. doi: 10.1016/j.avsg.2016.07.063. Epub 2016 Aug 13. PMID 27531079
- [Background] Newhall K, Suckow B, Spangler E, Brooke BS, Schanzer A, Tan TW, Burnette M, Edelen MO, Farber A, Goodney P; VAPOR investigators. Impact and Duration of Brief Surgeon-Delivered Smoking Cessation Advice on Attitudes Regarding Nicotine Dependence and Tobacco Harms for Patients with Peripheral Arterial Disease. Ann Vasc Surg. 2017 Jan;38:113-121. doi: 10.1016/j.avsg.2016.06.005. Epub 2016 Aug 10. PMID 27521828
- [Background] Chin JA, Skrip L, Sumpio BE, Cardella JA, Indes JE, Sarac TP, Dardik A, Ochoa Chaar CI. Percutaneous endovascular aneurysm repair in morbidly obese patients. J Vasc Surg. 2017 Mar;65(3):643-650.e1. doi: 10.1016/j.jvs.2016.06.115. Epub 2016 Dec 27. PMID 28034584
- [Background] Wang T, Shu C, Li M, Li QM, Li X, Qiu J, Fang K, Dardik A, Yang CZ. Thoracic Endovascular Aortic Repair With Single/Double Chimney Technique for Aortic Arch Pathologies. J Endovasc Ther. 2017 Jun;24(3):383-393. doi: 10.1177/1526602817698702. Epub 2017 Mar 21. PMID 28387611
- [Background] Wang T, Shu C, Li M, Dardik A, Li QM. In vitro Stent Graft Fenestration to Preserve All Supra-aortic Branches in the Treatment of a Stanford Type A Aortic Arch Dissection. Chin Med J (Engl). 2017 Aug 5;130(15):1878-1879. doi: 10.4103/0366-6999.211544. No abstract available. PMID 28748863
- [Background] Sadaghianloo N, Declemy S, Dardik A. Reply. J Vasc Surg. 2017 Mar;65(3):929-930. doi: 10.1016/j.jvs.2016.08.105. No abstract available. PMID 28236933
- [Background] Walsworth MK, de Bie R, Figoni SF, O'Connell JB. Peripheral Artery Disease: What You Need to Know. J Orthop Sports Phys Ther. 2017 Dec;47(12):957-964. doi: 10.2519/jospt.2017.7442. Epub 2017 Oct 9. PMID 28992768
- [Background] Archie M, Archie M, O'Connell J, DeRubertis BG. Underutilization of Thrombolytic Therapy for Patients Diagnosed with Acute Deep Venous Thrombosis in the Outpatient Setting. Ann Vasc Surg. 2018 May;49:255-260. doi: 10.1016/j.avsg.2018.02.005. Epub 2018 Feb 28. PMID 29499353
- [Background] Gelabert HA, Rigberg DA, O'Connell JB, Jabori S, Jimenez JC, Farley S. Transaxillary decompression of thoracic outlet syndrome patients presenting with cervical ribs. J Vasc Surg. 2018 Oct;68(4):1143-1149. doi: 10.1016/j.jvs.2018.01.057. Epub 2018 Apr 25. PMID 29705086
- [Background] Brooke BS, Slager SL, Swords DS, Weir CR. Patient and caregiver perspectives on care coordination during transitions of surgical care. Transl Behav Med. 2018 May 23;8(3):429-438. doi: 10.1093/tbm/ibx077. PMID 29800402
- [Background] Kim JJ, Mills JL, Braun J, Barshes N, Kougias P, Younes HK. Arteriovenous fistula maturation rate is not affected by ipsilateral tunneled dialysis catheter. J Vasc Surg. 2019 Nov;70(5):1629-1633. doi: 10.1016/j.jvs.2019.01.084. Epub 2019 Jun 21. PMID 31230847
- [Background] Anderson PB, Wanken ZJ, Perri JL, Columbo JA, Kang R, Spangler EL, Newhall K, Brooke BS, Dosluoglu H, Lee ES, Raffetto JD, Henke PK, Tang GL, Mureebe L, Kougias P, Johanning J, Arya S, Scali ST, Stone DH, Suckow BD, Orion K, Halpern V, O'Connell J, Inhat D, Nelson P, Tzeng E, Zhou W, Barry M, Sirovich B, Goodney PP; PROVE-AAA Study Team. Patient information sources when facing repair of abdominal aortic aneurysm. J Vasc Surg. 2020 Feb;71(2):497-504. doi: 10.1016/j.jvs.2019.04.460. Epub 2019 Jul 26. PMID 31353272
- [Background] Columbo JA, Kang R, Spangler EL, Newhall K, Brooke BS, Dosluoglu H, Lee ES, Raffetto JD, Henke PK, Tang GS, Mureebe L, Kougias P, Johanning J, Arya S, Scali ST, Stone DH, Suckow BD, Orion K, Halpern V, O'Connell J, Inhat D, Nelson P, Tzeng E, Zhou W, Barry M, Sirovich B, Goodney PP; PROVE-AAA Study Team. Design of the PReferences for Open Versus Endovascular Repair of Abdominal Aortic Aneurysm (PROVE-AAA) Trial. Ann Vasc Surg. 2020 May;65:247-253. doi: 10.1016/j.avsg.2019.02.034. Epub 2019 May 8. PMID 31075459
- [Background] Tran HA, O'Connell JB, Lee UK, Polanco JC, Chang TI, Friedlander AH. Relationship between symptomatic lower limb peripheral artery disease and calcified carotid artery plaque detected on panoramic images of neurologically asymptomatic males. Dentomaxillofac Radiol. 2019 Jul;48(5):20180432. doi: 10.1259/dmfr.20180432. Epub 2019 Mar 19. PMID 30875245
- [Result] Fereydooni A, Nassiri N. Evaluation and management of the lateral marginal vein in Klippel-Trenaunay and other PIK3CA-related overgrowth syndromes. J Vasc Surg Venous Lymphat Disord. 2020 May;8(3):482-493. doi: 10.1016/j.jvsv.2019.12.003. Epub 2020 Feb 20. PMID 32089498
- [Result] Brahmandam A, Gholitabar N, Cardella J, Nassiri N, Dardik A, Georgi M, Ochoa Chaar CI. Discrepancy in Outcomes after Revascularization for Chronic Limb-Threatening Ischemia Warrants Separate Reporting of Rest Pain and Tissue Loss. Ann Vasc Surg. 2021 Jan;70:237-244. doi: 10.1016/j.avsg.2020.06.057. Epub 2020 Jul 10. PMID 32659417
- [Result] Bellamkonda KS, Yousef S, Nassiri N, Dardik A, Guzman RJ, Geirsson A, Ochoa Chaar CI. Trends and outcomes of thoracic endovascular aortic repair with open concomitant cervical debranching. J Vasc Surg. 2021 Apr;73(4):1205-1212.e3. doi: 10.1016/j.jvs.2020.07.103. Epub 2020 Aug 27. PMID 32861861
- [Result] Holeman TA, Peacock J, Beckstrom JL, Brooke BS. Patient-Surgeon Agreement in Assessment of Frailty, Physical Function, & Social Activity. J Surg Res. 2020 Dec;256:368-373. doi: 10.1016/j.jss.2020.06.059. Epub 2020 Jul 30. PMID 32739620
- [Result] DeAngelo MM, Peacock JB, Holeman TA, Maloney M, Beckstrom J, Brooke BS. Long-Term Functional Decline Following Vascular Surgery Among Vulnerable Adults. Ann Vasc Surg. 2021 Oct;76:87-94. doi: 10.1016/j.avsg.2021.04.002. Epub 2021 Apr 22. PMID 33895257
- [Result] Eid MA, Barnes JA, Mehta K, Wanken Z, Columbo J, Kang R, Newhall K, Halpern V, Raffetto J, Kougias P, Henke P, Tang G, Mureebe L, Johanning J, Tzeng E, Scali S, Stone D, Suckow B, Lee E, Arya S, Orion K, O'Connell J, Brooke B, Ihnat D, Dosluoglu H, Zhou W, Nelson P, Spangler E, Barry M, Sirovich B, Goodney P. Factors associated with preference of choice of aortic aneurysm repair in the PReference for Open Versus Endovascular repair of AAA (PROVE-AAA) study. J Vasc Surg. 2022 Dec;76(6):1556-1564. doi: 10.1016/j.jvs.2022.06.018. Epub 2022 Jul 19. PMID 35863555
- [Derived] Eid MA, Barry MJ, Tang GL, Henke PK, Johanning JM, Tzeng E, Scali ST, Stone DH, Suckow BD, Lee ES, Arya S, Brooke BS, Nelson PR, Spangler EL, Murebee L, Dosluoglu HH, Raffetto JD, Kougais P, Brewster LP, Alabi O, Dardik A, Halpern VJ, O'Connell JB, Ihnat DM, Zhou W, Sirovich BE, Metha K, Moore KO, Voorhees A, Goodney PP; Preferences for Open Versus Endovascular Repair of Abdominal Aortic Aneurysm (PROVE-AAA) Study Team. Effect of a Decision Aid on Agreement Between Patient Preferences and Repair Type for Abdominal Aortic Aneurysm: A Randomized Clinical Trial. JAMA Surg. 2022 Sep 1;157(9):e222935. doi: 10.1001/jamasurg.2022.2935. Epub 2022 Sep 14. PMID 35947375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study we had 241 total enrollments, including three dual enrollments. Three participants were enrolled at one Prove-AAA site and were then subsequently enrolled at another Prove-AAA site. All three of these participants were fully withdrawn via a protocol deviation filed with the central institutional review board to only be enrolled at one site. Out of the 238 enrolled participants three were fully withdrawn via protocol deviation.
Units Other Than Participants: Study Sites
Groups:
- Veteran's Hospital Vascular Surgery Clinics Using Decision Aid: Participants in this arm of the study were given a information packet describing endovascular repair and Open AAA surgery prior to seeing their vascular surgeon.
- Veterans Hospital Vascular Surgery Clinics Providing Usual Care: Participants in this arm of the study did not receive an informational packet prior to visiting with their vascular surgeon
Period: Overall Study
Arm/Group | Veteran's Hospital Vascular Surgery Clinics Using Decision Aid | Veterans Hospital Vascular Surgery Clinics Providing Usual Care
Started | 126; 11 Study Sites (2 participants in this group were withdrawn because they were found later to not meet enrollment criteria.) | 109; 11 Study Sites (1 participant in this group was withdrawn because they were found later to not meet enrollment criteria.)
Completed | 95; 11 Study Sites | 87; 11 Study Sites
Not Completed | 31; 0 Study Sites | 22; 0 Study Sites
Not completed — Did not have AAA surgery | 28 | 15
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participations reflects the Number of Participations who started the study as described in the Participant Flow, Overall Study Table.
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | Control | Total
Number analyzed (Participants) | 126 | 109 | 235
Age, Continuous [Mean (Full Range); unit: years] | 73 [66 to 80] | 74 [66 to 82] | 74 [66 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 126 | 108 | 234
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 111 | 97 | 208
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Veteran Preference for Repair Type
Description: The investigators' survey will measure the effect of the decision aid on Veterans preference for repair type for abdominal aortic aneurysms and domains associated with preference for each repair type (endovascular or open)
Time Frame: 30 days
Population: These numbers differ from the participant flow module due to omitted survey answers by participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Control
Number analyzed (Participants) | 120 | 105
Participants
  Veteran Preference for Open | 25 | 25
  Veteran Preference for EVAR | 95 | 80

2. Primary Outcome: Agreement Between Veterans Preferences for Repair Type and Actual Repair Type
Description: The investigators' survey instruments will assess the effect of the decision aid on the agreement between Veteran's preference for repair type and actual repair type they receive
Time Frame: 30 days
Population: These numbers differ from the participant flow module because only 98 participants received AAA repair in the intervention group and 94 in the control group received AAA repair. From these participants who had AAA repair, analysis was limited to 94 in the decision aid group and 90 in the control group due to participants being lost to follow-up or omitted survey answers.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Control
Number analyzed (Participants) | 94 | 90
Participants
  Veterans that had agreement between preference and repair received | 88 | 75
  Veterans that did not have agreement between preference and repair received | 6 | 15

3. Secondary Outcome: Decision Regret Scale
Description: The investigators will use the patient satisfaction questionnaire short form 18 to assess patient satisfaction. Patient satisfaction will be reported based on the average Decision Process Score for both decision and control groups, with a score of 5 representing the highest level of satisfaction and a score of 0 representing the lowest level of satisfaction.
Time Frame: 30 days
Population: These numbers differ from the participant flow module due to omitted survey answers by participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Decision Aid | Control
Number analyzed (Participants) | 125 | 107
score on a scale | 4.9 [3.2 to 5.4] | 4.95 [2.9 to 5.6]

ADVERSE EVENTS:
Time Frame: Each subject was followed from the time of enrollment for two years, or until AAA repair occurred.
Description: The investigators only recorded mortality prior to study completion (prior to Post- Surgery PSQ) as an adverse event. All deaths are not related to study participation, this study involved answering surveys and no medical intervention was involved.
Arm/Group | Decision Aid | Control
All-Cause Mortality (participants affected / at risk) | 8/126 | 5/109
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/109
Other Adverse Events (participants affected / at risk) | 0/126 | 0/109

LIMITATIONS AND CAVEATS:
While decision aids for patients facing aortic aneurysm repair are associated with better alignment between preferences and outcomes, use of a decision aid may add time required for clinic visits in real-world practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03115346/Prot_SAP_001.pdf